CLINICAL TRIAL: NCT01645956
Title: Consistency in Individual Differences in Energy Intake Following Acute Exercise
Status: Completed | Type: Observational
Sponsor: The Miriam Hospital (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Other Study IDs: 400012; 1R03CA162965-01A1 (NIH)
Record Dates: First submitted 2012-07-18; First posted 2012-07-20 (Estimated); Last update posted 2015-02-19 (Estimated); Status verified 2012-07

CONDITIONS: Obesity; Sedentary
Keywords: obesity; exercise; energy intake; physical activity
MeSH Terms: conditions — Obesity; Sedentary Behavior; Motor Activity

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Single group

SUMMARY:
The importance of exercise for weight control is well documented; however if exercise results in an increase in food intake, the beneficial effect of exercise may not be seen. This study addresses a gap in the current literature and examines why some people eat more after exercise and why some people eat less and also examines whether these responses are consistent over time. Participants in this study will be asked to come to our center on 7 different occasions over a 3-4 month period. The first visit will be an assessment visit where body weight and body composition will be measured, questionnaires will be completed, and an exercise test will be performed. During the remaining 6 visits (3 pairs of sessions with visits in each pair separated by 48-96 hours) the procedures will be nearly identical. Upon arrival at our center, participants will consume a meal replacement, complete a series of questionnaires and then either rest or walk on a treadmill for 30 minutes (3 days will be resting and 3 will be exercising). One hour following the exercise/resting session, individuals will be given access to a buffet of food, unaware that their food intake will be monitored. All food will be weighed and measured before and after the eating period and the amount of food consumed after each pair of exercise and resting conditions will be compared to one another. It is hypothesized that the difference in food intake will be consistent across pairs of testing sessions. Findings from this study will help us to better understand the relationship between exercise and food intake and may ultimately lead to future studies that can address the clinically significant question of why some individuals gain weight and others lose weight when engaging in exercise training programs. Findings from this study may also help to develop exercise programs that maximize the beneficial effect of exercise on body weight.

ELIGIBILITY:
Inclusion Criteria:

* Age 18-45 years
* BMI between 25.0 and <35.0 kg/m2
* Female
* Sedentary, defined as exercising at a moderate-intensity for less than 60 minutes/week over the past 6 months.

Exclusion Criteria:

* Presence of any condition that would limit one's ability from exercising (i.e., orthopedic limitations)
* Recent weight gain or weight loss (± 10 pounds within the past 6 months)
* Currently enrolled in a weight loss program
* History of heart disease or diabetes
* Currently taking any medication that would alter heart rate (e.g., beta blocker) or metabolism
* Women who are pregnant, planning on becoming pregnant in the next 2 months, or those pregnant within the past 6 months
* Uncontrolled hypertension (currently taking blood pressure medication or having a resting systolic blood pressure ≥140/90 mmHg
* Get an average of <6 hours of sleep/night
* Does not currently eat breakfast regularly
* Known food allergies to test foods or states a disliking or unwillingness to eat more than 25% of the buffet foods.

Ages: 18 Years to 45 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Study Population: Relatively sedentary (exercising less than 60 minutes/week over the past 6 months) overweight and obese (BMI: 25.0 to <35.0 kg/m2) women between the ages of 18 and 45.
Sampling Method: Non-Probability Sample
Enrollment: 28 (Actual)
Dates: Start 2012-07; Primary Completion 2014-07 (Actual); Study Completion 2014-07 (Actual)

PRIMARY OUTCOMES:
energy intake | 1 hour post exercise/rest

CONTACTS AND LOCATIONS:
Overall Officials: Jessica L Unick, PhD, Principal Investigator — The Miriam Hospital
Locations (1):
- Weight Control and Diabetes Research Center, Providence, Rhode Island, United States